CLINICAL TRIAL: NCT00257244
Title: Inflammation and the Host Response to Injury
Brief Title: Inflammation and the Host Response to Injury (Burns)
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ronald G. Tompkins, Chief, Burns Service, Massachusetts General Hospital
Other Study IDs: 2 U54 GM062119_burn; U54GM062119 (NIH)
Record Dates: First submitted 2005-11-18; First posted 2005-11-22 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Trauma; Burns; Multiple Organ Failure
Keywords: Immunity, innate; Inflammation; Genomics; Proteomics
MeSH Terms: conditions — Wounds and Injuries; Burns; Multiple Organ Failure; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, blood leukocyte nucleic acids (RNA), solid tissue nucleic acids (only RNA, no DNA)
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to help improve our understanding of the biology involved in the body's response to serious trauma or burn injury. The host response to trauma and burns is a collection of physiological and pathophysiological processes that depend critically upon the regulation of the human innate immune system, with particular emphasis on the inflammatory component of that system. No single research center or small group of centers has the capacity to delineate the integrated response of this complex biological system, which involves multiple molecular and genetic interactions that vary in time. Our proposal promotes the identification of important dynamic relationships that regulate the integration of this complex biological system, with the expectation that this understanding will ultimately impact the diagnosis, prognosis, and treatment of the hospitalized, severely injured patient.

DETAILED DESCRIPTION:
This large-scale collaborative project provides the means to acquire the necessary new knowledge directly in humans. Knowledge will be acquired using diverse state-of-the-art genomic and proteomic technologies, a highly complex clinical, proteomic, and genomic database, as well as newly-developed, novel analytical tools to probe this complex dataset. Our analytical capabilities at the genomic and proteomic level are now rapidly evolving and our ability to link these genomic and proteomic data to pathways and functional modules will help us more closely link this cellular data to immunological processes and ultimately, to the phenotypic response (i.e., trajectory) in the injured host. As a result, potential interventions, whether through our Program or other funding mechanisms, can be more effectively designed.

ELIGIBILITY:
Inclusion Criteria:

* Burn patients of all ages with 20% or greater of total body surface area burns that require surgical treatment
* Burn patients admitted to the burn unit within 96 hours (4 days) of burn injury

All patients meeting these criteria are entered into the epidemiologic database and assessed for specific exclusion criteria to establish whether serial blood draws are warranted.

Exclusion Criteria:

* Injury caused by chemical agent
* Deep injury caused by conduction of electrical current or charge
* Decision not to treat due to severity of injury
* Anoxic brain injury that is not expected to result in complete recovery
* Associated multiple injuries exclusive of burns (ISS >=25)
* Pre-morbid condition: Severe congestive heart failure (measured ejection fraction <20%)
* Pre-morbid condition: Malignancy currently under treatment
* Pre-morbid condition: Medical condition requiring systemic glucocorticoid treatment
* Pre-morbid condition: current systemic immunosuppression for organ transplant or chronic inflammatory condition

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Acute hospitalized burn patients
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2004-04; Primary Completion 2013-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Time to death | Within two years of burn injury
Change in gene expression after burn injury | Up to two years after burn injury
Number and type of complications | Up to two years after burn injury

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G. Tompkins, MD, ScD, Principal Investigator — Massachusetts General Hospital
Locations (4):
- United States (4):
  - Loyola University Medical Center at Loyola in Chicago, Maywood, Illinois
  - Southwestern Medical Center at University of Texas Southwestern, Dallas, Texas
  - University of Texas at Galveston-Shriners Burn Hospital- Galveston, Galveston, Texas
  - Harborview Medical Center at University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Curated and validated data are available to Consortium Members

REFERENCES:
- [Background] Brownstein BH, Logvinenko T, Lederer JA, Cobb JP, Hubbard WJ, Chaudry IH, Remick DG, Baker HV, Xiao W, Mannick JA. Commonality and differences in leukocyte gene expression patterns among three models of inflammation and injury. Physiol Genomics. 2006 Feb 14;24(3):298-309. doi: 10.1152/physiolgenomics.00213.2005. Epub 2005 Dec 20. PMID 16478828
- [Background] Silver GM, Klein MB, Herndon DN, Gamelli RL, Gibran NS, Altstein L, McDonald-Smith GP, Tompkins RG, Hunt JL; Inflammation and the Host Response to Trauma, Collaborative Research Program. Standard operating procedures for the clinical management of patients enrolled in a prospective study of Inflammation and the Host Response to Thermal Injury. J Burn Care Res. 2007 Mar-Apr;28(2):222-30. doi: 10.1097/BCR.0B013E318031AA44. PMID 17351437
- [Background] Lederer JA, Brownstein BH, Lopez MC, Macmillan S, Delisle AJ, Macconmara MP, Choudhry MA, Xiao W, Lekousi S, Cobb JP, Baker HV, Mannick JA, Chaudry IH; Inflammation and the Host Response to Injury Collaborative Research Program Participants. Comparison of longitudinal leukocyte gene expression after burn injury or trauma-hemorrhage in mice. Physiol Genomics. 2008 Feb 19;32(3):299-310. doi: 10.1152/physiolgenomics.00086.2007. Epub 2007 Nov 6. PMID 17986522
- [Result] Klein MB, Silver G, Gamelli RL, Gibran NS, Herndon DN, Hunt JL, Tompkins RG; Inflammation and the Host Response to Injury Investigators. Inflammation and the host response to injury: an overview of the multicenter study of the genomic and proteomic response to burn injury. J Burn Care Res. 2006 Jul-Aug;27(4):448-51. doi: 10.1097/01.BCR.0000227477.33877.E6. PMID 16819346
- [Result] Klein MB, Hayden D, Elson C, Nathens AB, Gamelli RL, Gibran NS, Herndon DN, Arnoldo B, Silver G, Schoenfeld D, Tompkins RG. The association between fluid administration and outcome following major burn: a multicenter study. Ann Surg. 2007 Apr;245(4):622-8. doi: 10.1097/01.sla.0000252572.50684.49. PMID 17414612
- [Result] Russom A, Sethu P, Irimia D, Mindrinos MN, Calvano SE, Garcia I, Finnerty C, Tannahill C, Abouhamze A, Wilhelmy J, Lopez MC, Baker HV, Herndon DN, Lowry SF, Maier RV, Davis RW, Moldawer LL, Tompkins RG, Toner M; Inflammation and Host Response to Injury Large Scale Collaborative Research Program. Microfluidic leukocyte isolation for gene expression analysis in critically ill hospitalized patients. Clin Chem. 2008 May;54(5):891-900. doi: 10.1373/clinchem.2007.099150. Epub 2008 Mar 28. PMID 18375483
- [Result] Kotz KT, Xiao W, Miller-Graziano C, Qian WJ, Russom A, Warner EA, Moldawer LL, De A, Bankey PE, Petritis BO, Camp DG 2nd, Rosenbach AE, Goverman J, Fagan SP, Brownstein BH, Irimia D, Xu W, Wilhelmy J, Mindrinos MN, Smith RD, Davis RW, Tompkins RG, Toner M; Inflammation and the Host Response to Injury Collaborative Research Program. Clinical microfluidics for neutrophil genomics and proteomics. Nat Med. 2010 Sep;16(9):1042-7. doi: 10.1038/nm.2205. Epub 2010 Aug 29. PMID 20802500
- [Result] Xiao W, Mindrinos MN, Seok J, Cuschieri J, Cuenca AG, Gao H, Hayden DL, Hennessy L, Moore EE, Minei JP, Bankey PE, Johnson JL, Sperry J, Nathens AB, Billiar TR, West MA, Brownstein BH, Mason PH, Baker HV, Finnerty CC, Jeschke MG, Lopez MC, Klein MB, Gamelli RL, Gibran NS, Arnoldo B, Xu W, Zhang Y, Calvano SE, McDonald-Smith GP, Schoenfeld DA, Storey JD, Cobb JP, Warren HS, Moldawer LL, Herndon DN, Lowry SF, Maier RV, Davis RW, Tompkins RG; Inflammation and Host Response to Injury Large-Scale Collaborative Research Program. A genomic storm in critically injured humans. J Exp Med. 2011 Dec 19;208(13):2581-90. doi: 10.1084/jem.20111354. Epub 2011 Nov 21. PMID 22110166
- [Result] Finnerty CC, Jeschke MG, Herndon DN, Gamelli R, Gibran N, Klein M, Silver G, Arnoldo B, Remick D, Tompkins RG; Investigators of the Inflammation and the Host Response Glue Grant. Temporal cytokine profiles in severely burned patients: a comparison of adults and children. Mol Med. 2008 Sep-Oct;14(9-10):553-60. doi: 10.2119/2007-00132.Finnerty. PMID 18548133
- [Result] Qian WJ, Liu T, Petyuk VA, Gritsenko MA, Petritis BO, Polpitiya AD, Kaushal A, Xiao W, Finnerty CC, Jeschke MG, Jaitly N, Monroe ME, Moore RJ, Moldawer LL, Davis RW, Tompkins RG, Herndon DN, Camp DG, Smith RD; Inflammation and the Host Response to Injury Large Scale Collaborative Research Program. Large-scale multiplexed quantitative discovery proteomics enabled by the use of an (18)O-labeled "universal" reference sample. J Proteome Res. 2009 Jan;8(1):290-9. doi: 10.1021/pr800467r. PMID 19053531
- [Result] Qian WJ, Petritis BO, Kaushal A, Finnerty CC, Jeschke MG, Monroe ME, Moore RJ, Schepmoes AA, Xiao W, Moldawer LL, Davis RW, Tompkins RG, Herndon DN, Camp DG 2nd, Smith RD; Inflammation and the Host Response to Injury Large Scale Collaborative Research Program. Plasma proteome response to severe burn injury revealed by 18O-labeled "universal" reference-based quantitative proteomics. J Proteome Res. 2010 Sep 3;9(9):4779-89. doi: 10.1021/pr1005026. PMID 20698492
- [Result] Jeschke MG, Finnerty CC, Herndon DN, Song J, Boehning D, Tompkins RG, Baker HV, Gauglitz GG. Severe injury is associated with insulin resistance, endoplasmic reticulum stress response, and unfolded protein response. Ann Surg. 2012 Feb;255(2):370-8. doi: 10.1097/SLA.0b013e31823e76e7. PMID 22241293
- [Result] Seok J, Warren HS, Cuenca AG, Mindrinos MN, Baker HV, Xu W, Richards DR, McDonald-Smith GP, Gao H, Hennessy L, Finnerty CC, Lopez CM, Honari S, Moore EE, Minei JP, Cuschieri J, Bankey PE, Johnson JL, Sperry J, Nathens AB, Billiar TR, West MA, Jeschke MG, Klein MB, Gamelli RL, Gibran NS, Brownstein BH, Miller-Graziano C, Calvano SE, Mason PH, Cobb JP, Rahme LG, Lowry SF, Maier RV, Moldawer LL, Herndon DN, Davis RW, Xiao W, Tompkins RG; Inflammation and Host Response to Injury, Large Scale Collaborative Research Program. Genomic responses in mouse models poorly mimic human inflammatory diseases. Proc Natl Acad Sci U S A. 2013 Feb 26;110(9):3507-12. doi: 10.1073/pnas.1222878110. Epub 2013 Feb 11. PMID 23401516
- [Result] Finnerty CC, Jeschke MG, Qian WJ, Kaushal A, Xiao W, Liu T, Gritsenko MA, Moore RJ, Camp DG 2nd, Moldawer LL, Elson C, Schoenfeld D, Gamelli R, Gibran N, Klein M, Arnoldo B, Remick D, Smith RD, Davis R, Tompkins RG, Herndon DN; Investigators of the Inflammation and the Host Response Glue Grant. Determination of burn patient outcome by large-scale quantitative discovery proteomics. Crit Care Med. 2013 Jun;41(6):1421-34. doi: 10.1097/CCM.0b013e31827c072e. PMID 23507713
- [Result] Warren HS, Tompkins RG, Mindrinos MN, Xiao W, Davis RW. Reply to Cauwels et al.: Of men, not mice, and inflammation. Proc Natl Acad Sci U S A. 2013 Aug 20;110(34):E3151. doi: 10.1073/pnas.1308943110. No abstract available. PMID 24137663
- [Result] Jeschke MG, Finnerty CC, Emdad F, Rivero HG, Kraft R, Williams FN, Gamelli RL, Gibran NS, Klein MB, Arnoldo BD, Tompkins RG, Herndon DN. Mild obesity is protective after severe burn injury. Ann Surg. 2013 Dec;258(6):1119-29. doi: 10.1097/SLA.0b013e3182984d19. PMID 23877367
- [Result] Klein MB, Goverman J, Hayden DL, Fagan SP, McDonald-Smith GP, Alexander AK, Gamelli RL, Gibran NS, Finnerty CC, Jeschke MG, Arnoldo B, Wispelwey B, Mindrinos MN, Xiao W, Honari SE, Mason PH, Schoenfeld DA, Herndon DN, Tompkins RG; Inflammation and Host Response to Injury, and Large-Scale Collaborative Research Program. Benchmarking outcomes in the critically injured burn patient. Ann Surg. 2014 May;259(5):833-41. doi: 10.1097/SLA.0000000000000438. PMID 24722222
- [Result] Tompkins RG. Survival from burns in the new millennium: 70 years' experience from a single institution. Ann Surg. 2015 Feb;261(2):263-8. doi: 10.1097/SLA.0000000000000623. PMID 24670865
- [Result] Warren HS, Tompkins RG, Moldawer LL, Seok J, Xu W, Mindrinos MN, Maier RV, Xiao W, Davis RW. Mice are not men. Proc Natl Acad Sci U S A. 2015 Jan 27;112(4):E345. doi: 10.1073/pnas.1414857111. Epub 2014 Dec 24. No abstract available. PMID 25540422
- See also: Information about the study and its goals. Contains links to study related publications, resources, and participating institutions — http://www.gluegrant.org/